CLINICAL TRIAL: NCT00920829
Title: Genetic and Brain Mechanisms of Naltrexone?s Treatment Efficacy for Alcoholism
Brief Title: Genetic and Brain Mechanisms of Naltrexone's Treatment Efficacy for Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ANTON-1R01AA017633-01A1
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence; Alcoholism; Naltrexone; Substance Abuse; Genetics
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A118G A/A with Naltrexone (Active Comparator): Individuals with the OPRM1 genotype Asn40 are given naltrexone 50 mg after 2 days at 25 mg for 16 weeks with Medication Management 9 visits in 16 weeks
  Interventions: Drug: Naltrexone 50 Mg
- A118G A/A with Placebo (Placebo Comparator): Individuals with the OPRM1 genotype Asn40 are given Placebo for 16 weeks with Medication Management in 16 weeks
  Interventions: Drug: Placebo
- A118G Any G with Naltrexone (Active Comparator): Individuals with the OPRM1 genotype Any G (Asp) are given naltrexone 50 mg after 2 days of naltrexone 25 mg for 16 weeks with Medication Management 9 visits in 16 weeks
  Interventions: Drug: Naltrexone 50 Mg
- A118G Any G with Placebo (Placebo Comparator): Individuals with the OPRM1 genotype Any G (Asp) are given 50 mg naltrexone after 2 days at 25 mg for 16 weeks with Medication Management 9 visits in 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone 50 Mg — Naltrexone 25 or 50 mg per titration schedule
  Arms: A118G A/A with Naltrexone; A118G Any G with Naltrexone
Drug: Placebo — placebo
  Arms: A118G A/A with Placebo; A118G Any G with Placebo

SUMMARY:
The overarching aim of this trial is to evaluate naltrexone's efficacy in light of genetic variation and brain response to alcohol cues utilizing a neuroimaging paradigm. This trial has four specific aims. First, this trial will evaluate whether the presence of the OPRM1 Asp40 allele substitution is associated with improved treatment response to naltrexone in treatment-seeking alcoholics. Second, it will evaluate whether there is a difference in the naltrexone dampening of the alcohol cue-induced brain activation dependent on OPRM1 genotype. Third, it will explore whether alcohol cue-induced brain activation dampening by naltrexone might be a mediating factor in the treatment effects of naltrexone, the OPRM1 gene, or their interaction that might be observed in the first aim. Finally, this trial will evaluate the effect of medication compliance, or adverse effects, on the observed medication by genotype treatment response. A secondary aim will measure medication compliance and side effects based on OPRM1 genotype.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 70
2. Subjects will meet criteria for primary alcohol dependence
3. Consumes, on average, at least 5 standard drinks per day for men and 4 drinks per day for women in the 90 days pre-screening. Has at least 50% of days as heavy drinking days (as defined above).
4. Able to maintain sobriety for four days (with or without the aid of alcohol detoxification medications) as determined by self report and breathalyzer measurements
5. Able to read and understand questionnaires and informed consent
6. Lives within approximately 50 miles of the study site

Exclusion Criteria

1. Currently meets DSM IV criteria for any other psychoactive substance dependence disorder except nicotine dependence
2. Any psychoactive substance abuse, except marijuana, nicotine, and cocaine, within the last 30 days as evidenced by subject report, collateral report, or urine drug screen. May meet cocaine abuse criteria, but not dependence, and also must have two sequential urines free of illicit substances
3. Meets DSM IV criteria for current and active axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, or any other psychotic disorder or organic mental disorder
4. Meets DSM IV current criteria for dissociative disorder or eating disorders
5. Has current suicidal ideation or homicidal ideation
6. Need for maintenance or acute treatment with any psychoactive medication, except a stable dose (at least one month) of antidepressants
7. Need for maintenance on anti-seizure medications (including topiramate and gabapentin)
8. Use of disulfiram, acamprosate, or naltrexone in the last two weeks
9. Clinically significant medical problems such as cardiovascular, renal, GI, or endocrine problem that would impair participation or limit medication ingestion
10. Hepatocellular disease indicated by elevations of SGPT (ALT) and SGOT (AST) of at least 3.0 times normal at screening and/or after 5 days abstinence
11. Sexually active female of child-bearing potential who is pregnant (by urine HCG), nursing, or who is not willing to use a reliable form of birth control
12. Has current charges pending for a violent crime (not including DUI-related offenses)
13. Does not have a stable living situation
14. African American heritage due to low prevalence of Asp40 (also see Inclusion of Women and Minorities section)

Exclusion Criteria of fMRI Procedure

1. Having metal objects in the body that are deemed unsafe in the MRI environment.
2. Severe claustrophobia that cannot be managed with support and encouragement.
3. Morbid obesity such that placement in the MRI scanner is impossible.
4. History of significant head injury leading to unconsciousness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2009-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Anton, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Center for Drug and Alcohol Programs, Charleston, South Carolina
  - Medical University of South Carolin, Charleston, South Carolina

REFERENCES:
- [Result] Schacht JP, Randall PK, Latham PK, Voronin KE, Book SW, Myrick H, Anton RF. Predictors of Naltrexone Response in a Randomized Trial: Reward-Related Brain Activation, OPRM1 Genotype, and Smoking Status. Neuropsychopharmacology. 2017 Dec;42(13):2640-2653. doi: 10.1038/npp.2017.74. Epub 2017 Apr 14. PMID 28409564
- See also: Predictors of Naltrexone Response in a Randomized Trial: Reward-Related Brain Activation, OPRM1 Genotype, and Smoking Status. — https://www.ncbi.nlm.nih.gov/pubmed/28409564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 358 Subjects were recruited via media advertisements and clinical referrals and 355 provided a blood sample for A118G genotyping.
Pre-assignment Details: A118G genotyping was performed for 355 of these, 259 were A/A (Asn40) allele and 96 were any G (asp). Of the 259 Asn40 subjects, 89 were selected to participate 5 met exclusion criteria and 7 were lost or declined. Of the 96 Asp subjects, 9 met exclusion; 12 were lost or declined.
Groups:
- A118G A/A With Naltrexone: Individuals with the OPRM1 genotype Asn40 are given naltrexone 50 mg after 2 days at 25 mg for 16 weeks with Medication Management 9 visits in 16 weeks
  Naltrexone Hydrochloride 50 MG: Naltrexone 25 or 50 mg per tiration schedule
- A118G Any G With Naltrexone: Individuals with the OPRM1 genotype Any G (Asp) are given naltrexone 50 mg after 2 days of naltrexone 25 mg for 16 weeks with Medication Management 9 visits in 16 weeks
  Naltrexone Hydrochloride 50 MG: Naltrexone 25 or 50 mg per tiration schedule
Period: Allocation
Arm/Group | A118G A/A With Naltrexone | A118G A/A With Placebo | A118G Any G With Naltrexone | A118G Any G With Placebo
Started | 38 | 39 | 38 | 37
Completed | 35 | 38 | 38 | 35
Not Completed | 3 | 1 | 0 | 2
Not completed — No post randomization data | 3 | 1 | 0 | 2
Period: Available for Analysis
Arm/Group | A118G A/A With Naltrexone | A118G A/A With Placebo | A118G Any G With Naltrexone | A118G Any G With Placebo
Started | 35 | 38 | 38 | 35
Completed | 27 | 27 | 28 | 24
Not Completed | 8 | 11 | 10 | 11
Not completed — Withdrawal by Subject | 6 | 6 | 6 | 10
Not completed — Required Medical Treatment | 0 | 1 | 2 | 0
Not completed — Adverse Event | 1 | 2 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Required more treatment | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A118G A/A With Naltrexone | A118G A/A With Placebo | A118G Any G With Naltrexone | A118G Any G With Placebo | Total
Number analyzed (Participants) | 35 | 38 | 38 | 35 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (8.2) | 46.3 (10.8) | 50.3 (10.2) | 49.7 (10.6) | 49.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 13 | 11 | 45
  Male | 26 | 26 | 25 | 24 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 34 | 38 | 38 | 34 | 144
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Heavy Drinking Days by mu Opioid Receptor Gene
Time Frame: Time Line Follow-Back drinking collected at each of 9 visits (weeks 1, 2, 3, 4, 6, 8, 10, 12 and 16)
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | A118G A/A With Naltrexone | A118G A/A With Placebo | A118G Any G With Naltrexone | A118G Any G With Placebo
Number analyzed (Participants) | 35 | 38 | 38 | 35
percentage of days
  Month 1 | 11.0 (3.5) | 18.0 (3.4) | 11.8 (3.4) | 18.7 (3.6)
  Month 2 | 11.7 (4.5) | 25.8 (4.4) | 15.5 (4.4) | 19.7 (4.5)
  Month 3 | 10.4 (4.4) | 23.0 (4.3) | 16.9 (4.3) | 25.0 (4.4)
  Month 4 | 11.4 (4.7) | 18.1 (4.5) | 18.3 (4.5) | 28.7 (4.6)
Statistical Analysis 1: Comparison: A118G A/A With Naltrexone vs A118G A/A With Placebo vs A118G Any G With Naltrexone vs A118G Any G With Placebo; A linear mixed model with unstructured variance/covariance matrices was used to evaluate the primary outcome measure; Test type: Superiority; p = 0.724, Mixed Models Analysis
Statistical Analysis 2: Comparison: A118G A/A With Naltrexone vs A118G A/A With Placebo vs A118G Any G With Naltrexone vs A118G Any G With Placebo; This is a test of the main effect of medication, with a null hypothesis of no difference between Naltrexone and Placebo groups; Test type: Superiority; p = 0.023, Mixed Models Analysis

ADVERSE EVENTS:
Description: Number of subjects responding positively to queries in the SAFTEE instrument.
Groups:
- Placebo/ASN: ASN subjects given placebo
- Placebo/ASP: ASP subjects given placebo
- Naltrexone/ASN: ASN subjects given naltrexone
- Naltrexone/ASP: ASP subjects given naltrexone
Arm/Group | Placebo/ASN | Placebo/ASP | Naltrexone/ASN | Naltrexone/ASP
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35 | 0/35 | 1/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/35 | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 16/38 | 20/35 | 30/35 | 29/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/ASN (N=38) | Placebo/ASP (N=35) | Naltrexone/ASN (N=35) | Naltrexone/ASP (N=38)
Nausea (Gastrointestinal disorders) | 9 (9) | 9 (14) | 22 (27) | 13 (26)
Diarrhea (Gastrointestinal disorders) | 6 (8) | 9 (19) | 18 (28) | 16 (35)
abdominal pain (Gastrointestinal disorders) | 4 (6) | 5 (17) | 11 (22) | 16 (32)
dizziness (General disorders) | 6 (7) | 9 (21) | 14 (26) | 14 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No